CLINICAL TRIAL: NCT04210076
Title: Mindfulness Training for Small Teams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amishi Jha, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20191047; W81XWH1920064 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Change
Keywords: attentional performance; psychological well-being; operational performance
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Attention Training for Teams (MBAT-T) (Experimental): Teams randomized to this group will receive 4, 2-2.5-hour sessions delivered over 4 weeks of mindfulness training and 15 minutes of daily, out-of-class mindfulness exercises, that will be delivered and tracked using a measuring mindfulness application.
  Interventions: Behavioral: MBAT-T
- Mindfulness-Based Attention Training for Individuals (MBAT-I) (Active Comparator): Individuals randomized to this group will receive 4, 2-2.5-hour sessions delivered over 4 weeks of mindfulness training and 15 minutes of daily, out-of-class mindfulness exercises, that will be delivered and tracked using a measuring mindfulness application.
  Interventions: Behavioral: MBAT-I
- No-training (No Intervention): Teams will not engage in any mindfulness training

INTERVENTIONS:
Behavioral: MBAT-T — The MBAT-Team program builds on the basic 4-week, 8-hour MBAT-Soldier program. In addition to the basic program, MBAT-Team includes exercises promoting the cultivation of attention and emotion regulation in the service of effective team interactions (e.g., mindful communication and listening; monitoring and attention to the activities and emotional states of others, and additional practices to promote collective mindfulness).
  Arms: Mindfulness-Based Attention Training for Teams (MBAT-T)
Behavioral: MBAT-I — The MBAT-Individual program is based on the basic 4-week, 8-hour MBAT-Soldier curriculum.
  Arms: Mindfulness-Based Attention Training for Individuals (MBAT-I)

SUMMARY:
The purpose of this study is to look at how mindfulness training may influence how the participant thinks, feels, and acts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 18 and 65 years of age
* Individuals who are fluent English speakers
* Individuals who are active-duty service members
* Men and women of all races and ethnicities

Exclusion Criteria:

* Individuals who have a medical or neurological condition that might interfere with performance on the task in the study (e.g., epilepsy)
* Individuals with a history of hospitalization for psychological/mental health issues within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Change in Attentional Performance | Baseline (testing session 1) to week 5 (testing session 2)
  Attentional Performance as measured by the Sustained Attention Response Task (SART).This task uses a continuous performance paradigm involving button presses to frequently presented non-targets (numbers 1, 2, 4, 5, 6, 7, 8, and 9) but requires the participants to withhold their motor response to the infrequent target (number 3). Withholding responses only to infrequent targets encourages a pre-potent response and mind wandering. Real-time subjective experience of mind wandering during SART is assessed through experience-sampling probes randomly presented throughout the task.
Change in Working Memory Performance | Baseline (testing session 1) to week 5 (testing session 2)
  Working Memory Performance as measured by the Working memory task with Affective Distracters. In this task, participants are presented with a memory array that they are to encode and hold in memory during a delay interval. During the delay, emotionally negative or neutral scene images are presented.

SECONDARY OUTCOMES:
Change in Cohesion | Baseline (testing session 1) to week 5 (testing session 2)
  Cohesion as measured by 3 items adapted from a questionnaire developed by Podsakoff and MacKenzie. Scale items are rated on a scale from 1 to 5 (1 = strongly disagree, 5 = strongly agree), according to how much participants agree with each item.
Change in Team Situation Monitoring | Baseline (testing session 1) to week 5 (testing session 2)
  Team Situation Monitoring is measured by 7-item subscale of the Teamwork Perception Questionnaire, which assesses individuals' shared perceptions of group-level team skills and behavior. The scale consists of a list of items that are rated on a scale from 1 to 5 (1 = strongly disagree, 5 = strongly agree), according to how much participants agree with each item.
Change in Workgroup Emotional Intelligence | Baseline (testing session 1) to week 5 (testing session 2)
  Workgroup Emotional Intelligence as measured by the Workgroup Emotional Intelligence Profile, which is a 16-item measure of emotional intelligence abilities that manifest as behaviors in work teams. The scale consists of a list of items that are rated on a scale from 1 to 7 (1 = strongly disagree, 7 = strongly agree), according to how much participants agree with each item. This measure reflects an individual's judgment of their ability to monitor and manage their own emotions and the emotions of the members of their squad.
Change in Team Mindfulness | Baseline (testing session 1) to week 5 (testing session 2)
  Team Mindfulness as measured by the Team Mindfulness Scale, which is a 10-item scale measuring the individual's experience of their team interactions as mindful. The total score ranges from 1 to 5, with a higher score indicating an individual's perception of the team's attitudes and experiences as marked by greater mindfulness.
Change in Mindfulness | Baseline (testing session 1) to week 5 (testing session 2)
  Mindfulness as measured by the short version of the Five-Facet Mindfulness Questionnaire, which is a 15-item scale. The total score ranges from 15 to 75, with a higher score indicating greater levels of mindfulness in different aspects of one's life.
Change in Decentering | Baseline (testing session 1) to week 5 (testing session 2)
  Decentering as measured by the decentering sub-scale of the Experience Questionnaire, which is an 11-item scale measuring various thoughts and experiences, and the tendency to distance from those. The total score ranges from 1 to 55, with a higher score indicating higher levels of decentering.
Change in Psychological Health | Baseline (testing session 1) to week 5 (testing session 2)
  Psychological health as measured by the Patient Health Questionnaire, which is a 4-item scale measuring depression and anxiety. The total score ranges from 0 to 12, with higher scores indicating a higher level of depression and anxiety.
Change in Positive Affect | Baseline (testing session 1) to week 5 (testing session 2)
  Positive affect as measured by the short version of the Positive and Negative Affect Schedule (PANAS-10), a 5-item scale measuring the frequency of experiences of positive affect. The total score ranges from 5 to 25, with a higher score indicating a higher positive mood.
Change in Negative Affect | Baseline (testing session 1) to week 5 (testing session 2)
  Negative affect as measured by the short version of the Positive and Negative Affect Schedule (PANAS-10), a 5-item scale measuring the frequency of experiences of negative affect. The total score ranges from 5 to 25, with a higher score indicating a higher negative mood.
Change in Perceived Stress | Baseline (testing session 1) to week 5 (testing session 2)
  Perceived Stress as measured by the short version of the Perceived Stress Scale, which is a 4-item scale measuring the degree to which situations in one's life are viewed as stressful. The total score ranges from 0 to 16, with a higher score indicating higher levels of perceived stress.

OTHER OUTCOMES:
Change in Accuracy on Cognitive and Marksmanship Drills | Baseline (testing session 1) to week 5 (testing session 2)
  Marksmanship will be measured with drills involving synthetic rifles to interact with stimuli in an augmented reality environment. Accuracy in the drills will be scored from 0% to 100%, with a higher score indicating better performance.
Change in Reaction Time on Cognitive and Marksmanship Drills | Baseline (testing session 1) to week 5 (testing session 2)
  Marksmanship will be measured with drills involving synthetic rifles to interact with stimuli in an augmented reality environment. Reaction time will be measured in milliseconds, with lower values indicating faster responses.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi P Jha, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zanesco AP, Denkova E, Barry J, Jha AP. Mind wandering is associated with worsening attentional vigilance. J Exp Psychol Hum Percept Perform. 2024 Nov;50(11):1049-1066. doi: 10.1037/xhp0001233. Epub 2024 Aug 22. PMID 39172363